CLINICAL TRIAL: NCT06947863
Title: Comparison of the Clinical Effect on Common Low Back Pain of a Thermal Cure With Dry Rehabilitation: A Randomized Therapeutic Trial
Brief Title: Comparison of the Clinical Effect on Common Low Back Pain of a Thermal Cure With Dry Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Fazaa Alia, Associate professor, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONT-HMS
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: crenobalneotherapy; thermal cure; rehabilitation; randomized controlled trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The choice of the type of treatment to be delivered was determined by means of randomization provided by the senior investigator in accordance with the Zelen method. Neither the doctors participating in the study nor the patients were informed beforehand of the type of treatment that will be delivered, thermal cure (group 1) or dry rehabilitation (group 2).
  To calculate the number of subjects required in a group, we set alpha risk at 0.05, beta risk at 0.2 and the minimum difference of pain visual analog scale (VAS) to be highlighted between the 2 groups at 20 out of 100.
  To generate the randomization sequence, we randomly established a list of numbers using the EpiTable program in Epi Info (6.04d version), assigning treatment 1 to odd numbers and treatment 2 to even numbers. The number of patients was balanced after each 20-number sequence. Two groups of 37 patients each were formed. The patients were divided into 4 contingents.
Who Masked: Participant, Investigator
Masking Description: Neither the doctors participating in the study nor the patients were informed beforehand of the type of treatment that will be delivered, thermal cure (group 1) or dry rehabilitation (group 2).
  Each group of patients was unaware of the existence of the other group and its type of treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal cure (Active Comparator): The thermal treatment used hot, chlorinated and sodium water. Every day, the patients received 4 out of the 5 following treatments: underwater showers (15 minutes), shower-massage (10 minutes), hydromassage (20 minutes), swimming pool rehabilitation (20 minutes) and application of heated peloid (15 minutes).
  Patients were accommodated in the care center for 18 days. Treatments were delivered in the morning on a daily basis, except on Sundays.
  Interventions: Other: thermal cure
- dry rehabilitation (Active Comparator): The thermal treatment used hot, chlorinated and sodium water. Every day, the patients received 4 out of the 5 following treatments: underwater showers (15 minutes), shower-massage (10 minutes), hydromassage (20 minutes), swimming pool rehabilitation (20 minutes) and application of heated peloid (15 minutes).
  Interventions: Other: dry rehabilitation

INTERVENTIONS:
Other: thermal cure — The thermal treatment and physical rehabilitation therapy were administered at the same spa center of Jbal EL Ouest, situated to the west of the city of Zaghouan, 50 km from Tunis. Patients were accommodated in the care center for 18 days. Treatments were delivered in the morning on a daily basis, except on Sundays. The thermal treatment used hot, chlorinated and sodium water. Every day, the patients received 4 out of the 5 following treatments: underwater showers (15 minutes), shower-massage (10 minutes), hydromassage (20 minutes), swimming pool rehabilitation (20 minutes) and application of heated peloid (15 minutes).
  Arms: Thermal cure
Other: dry rehabilitation — The thermal treatment and physical rehabilitation therapy were administered at the same spa center of Jbal EL Ouest, situated to the west of the city of Zaghouan, 50 km from Tunis. Patients were accommodated in the care center for 18 days. Treatments were delivered in the morning on a daily basis, except on Sundays. The physical rehabilitation treatment was delivered in dry and included an analgesic physiotherapy based on electrotherapy (30 minutes) and muscle strengthening, as well as group rehabilitation.
  Other Names: physical rehabilitation
  Arms: dry rehabilitation

SUMMARY:
Objective: To compare the benefits, with regard to low back pain (LBP) symptoms, of a thermal cure and a dry rehabilitation treatment.

Methods: Randomized therapeutic trial including patients with LBP, randomly divided into two groups. Thermal cure consisted of underwater shower, massage-jet showers, hydro-massage, pool rehabilitation and peloid therapy. Dry rehabilitation consisted of analgesic physiotherapy, muscle strengthening and group physical rehabilitation. The primary endpoint was based on the Visual Analog Scale (VAS) of pain at day 18 (Day 18). The other outcome measures were the Oswestry Disability Index (ODI), the Short Form-36 (SF36) questionnaire and spine mobility. Follow-up was carried out for 12 months.

DETAILED DESCRIPTION:
Low back pain (LBP) is a very common pathology affecting more than 80% of the population. The pain and the limitation of movements cause significant functional discomfort, resulting in some form of disability and an added handicap. It therefore constitutes a major public health problem due to its impact on the quality of life and its high socio-economic cost.

The medical care for LBP aims to reduce pain and thus improve the functional capacities of patients. Among non-drug adjuvant treatments, the role of thermal cure is far from clear. Indeed, even if the use of thermo-mineral waters for therapeutic purposes is a very old and widespread practice in rheumatology, the study of the efficiency of thermal cures in the treatment of LBP, in particular compared to dry rehabilitation, has been the subject of only a limited number of medical publications. In Tunisia, the Tunisian Hydrotherapy Office estimates that at the end of 2017 the number of spa guests reached 51,324 for all the thermal resorts. However, there are no studies evaluating the effectiveness of such treatments.

We report the results of a randomized therapeutic trial, carried out with the aim of comparing the clinical effects of thermal cures and dry rehabilitation on common LBP.

Patient selection The selection of patients to be referred to the thermal center was made among patients treated in the rheumatology department of the Mongi Slim Hospital; a university hospital center located in La Marsa and not related to the thermal center. The inclusion visit allowed the investigating doctors to collect demographic data and clinical history, in order to verify the inclusion criteria and to have the informed consent signed in French or in Arabic depending on patients' choice.

Randomization The choice of the type of treatment to be delivered was determined by means of randomization provided by the senior investigator in accordance with the Zelen method. Neither the doctors participating in the study nor the patients were informed beforehand of the type of treatment that will be delivered, thermal cure (group 1) or dry rehabilitation (group 2). Each group of patients was unaware of the existence of the other group and its type of treatment.

To calculate the number of subjects required in a group, we set alpha risk at 0.05, beta risk at 0.2 and the minimum difference of pain VAS to be highlighted between the 2 groups at 20 out of 100.

To generate the randomization sequence, we randomly established a list of numbers using the EpiTable program in Epi Info (6.04d version), assigning treatment 1 to odd numbers and treatment 2 to even numbers. The number of patients was balanced after each 20-number sequence. Two groups of 37 patients each were formed. The patients were divided into 4 contingents.

Study protocol The thermal treatment and physical rehabilitation therapy were administered at the same spa center of Jbal EL Ouest, situated to the west of the city of Zaghouan, 50 km from Tunis. Patients were accommodated in the care center for 18 days. Treatments were delivered in the morning on a daily basis, except on Sundays. The thermal treatment used hot, chlorinated and sodium water. Every day, the patients received 4 out of the 5 following treatments: underwater showers (15 minutes), shower-massage (10 minutes), hydromassage (20 minutes), swimming pool rehabilitation (20 minutes) and application of heated peloid (15 minutes). The physical rehabilitation treatment was delivered in dry and included an analgesic physiotherapy based on electrotherapy (30 minutes) and muscle strengthening, as well as group rehabilitation.

Monitoring of care progress, compliance and tolerance during the treatment was carried out by the thermal center doctor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain (LBP) evolving for more than 12 weeks.
* Visual analog scale (VAS) of pain greater than 30.

Exclusion Criteria:

* Patients with a loss of autonomy or with impaired intellectual abilities
* Patients with contraindications to a thermal cure (infectious or progressive inflammatory pathologies, unbalanced blood hypertension, decompensated heart disease, respiratory failure, decompensated neurological or psychiatric illness, age greater than 75 years, pregnancy, purulent skin lesions).
* Patients having undergone an epidural infiltration (within 3 months) or spinal surgery (within 1 year)
* Patients who received physical rehabilitation or balneotherapy during the year preceding inclusion, and finally patients using stage 3 analgesics (World Health Organization classification).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
VAS pain | Day 18
  Pain was assessed using a visual analog scale (VAS) with a vertically held ruler graduated from 0 to 10. The VAS score for low back pain was then expressed in millimeters, ranging from 0 mm (no pain) to 100 mm (maximum pain). The primary endpoint was VAS pain, blindly assessed by the same doctor for each patient on the last day of the treatment (Day 18).

SECONDARY OUTCOMES:
VAS pain | at 3 months, 6 months and 12 months after the end of the treatment
  Pain was assessed using a visual analog scale (VAS) with a vertically held ruler graduated from 0 to 10. The VAS score for low back pain was then expressed in millimeters, ranging from 0 mm (no pain) to 100 mm (maximum pain). The secondary criteria were represented by the VAS pain at 3 months, 6 months and 12 months after the end of the treatment.
the OSWESTRY Disability Index (ODI) | at Day 18, month 3, month 6 and month 12.
  Functional capacity was assessed using the Oswestry Disability Index (ODI), for which the Arabic language version has been validated. It is a self-administered questionnaire consisting of eight items (pain, personal care, lifting, walking difficulties, sitting and standing positions, sleep, and social life). Each item includes six response options scored from 0 to 5. The total score is expressed as a percentage of disability, ranging from 0% (no disability) to 100% (total disability).
the quality of life score SF-36 | at Day 18, month 3, month 6 and month 12
  Patients' quality of life was assessed using the 36-Item Short Form Health Survey (SF-36), for which a validated Arabic version is available.The questionnaire includes 36 items assessing eight dimensions of quality of life: physical functioning, physical role limitations, bodily pain, general health, vitality, social functioning, emotional role limitations, and mental health. Each domain is scored from 0 to 100, with higher scores indicating better quality of life. The scores from the eight dimensions are used to calculate two summary scores: the Physical Component Summary (PCS), which includes physical functioning, physical role limitations, bodily pain, and general health; and the Mental Component Summary (MCS), which includes vitality, social functioning, emotional role limitations, and mental health.
spinal mobility | at Day 18, month 3, month 6 and month 12
  Assessment of Spinal Mobility The Schöber index assesses lumbar spine flexibility. It measures the distance between a horizontal landmark at the level of the L5 vertebra and a second landmark located 10 centimeters above it during maximal trunk flexion with feet together. A normal value is +5 cm.
  The fingertip-to-floor distance in forward flexion refers to the distance between the floor and the tip of the middle finger during maximal trunk flexion with feet together. The normal value is 0 cm.
  The fingertip-to-floor distance in lateral flexion is the difference between the fingertip-to-floor distance in the neutral position and that in lateral bending, with the iliac crest stabilized. It is expressed in centimeters.
  Inverse Schöber Index measures the distance between a horizontal landmark at the level of the L5 vertebra and a point 10 cm below it during maximal trunk extension

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Laatar, Professor, Study Chair — Rheumatology department, Mongi Slim Hospital, La Marsa, Tunisia; Alia Fazaa, Associate Professor, Principal Investigator — Rheumatology department, Mongi Slim Hospital, la Marsa, Tunisia
Locations (1):
- Mongi Slim Hospital, La Marsa, Sidi Daoued, Tunisia

IPD SHARING:
Plan to Share IPD: No